CLINICAL TRIAL: NCT06024759
Title: Long Term Registry of Patients With Left Ventricular Non-Compaction and Predictors of Adverse Outcomes
Brief Title: Predictors of Risk in Left Ventricular Non-Compaction
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 13529
Record Dates: First submitted 2023-07-31; First posted 2023-09-06 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Left Ventricular Noncompaction
Keywords: LVNC; Left Ventricular Non-Compaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: None Retained — Genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Individuals in this group were previously seen by physicians at the Inherited Arrhythmia Clinic at University Hospital, London Health Sciences Centre, yet are no longer being actively followed here anymore. These patients will have their data retrospectively obtained annually, ten years into the past, to collect data on key variables providing insight on LVNC progression over time.
- Prospective Cohort: Patients being actively followed up by physicians at the Inherited Arrhythmia Clinic will be approached either in person or via e-mail for consent and enrollment into this study. These patients will have their medical charts accessed annually to collect data on key variables providing insight on LVNC progression over time.

SUMMARY:
The goal of this study is to learn more about the risk factors associated with left ventricular non-compaction (LVNC) and the predictors of adverse outcomes associated with LVNC. The main questions this study aims to answer are as follows.

* Are there any genetic mutations that impact the risk of LVNC patients developing ventricular arrhythmias?
* Does LV myocardial strain increase risk stratification in the LVNC population with or without genetic mutations?
* What are some of the determinants that cause LV dysfunction in LVNC?
* What are other risk stratifiers (ex. premature ventricular contraction (PVC) burden on Holter, non-sustained ventricular tachycardia (NSVT) on stress test) that lead to an outcome of ICD implantation?

Participants will have their medical records accessed annually for a span of ten years, either prospectively or retrospectively depending on whether they are being actively followed by physicians at the Inherited Arrhythmia Clinic or not, to evaluate LVNC progression over time. This data will be stored in a large clinical registry with the London Heart Rhythm Program at the London Health Sciences Centre, University Hospital Campus.

DETAILED DESCRIPTION:
Left ventricular noncompaction (LVNC) is a congenital cardiomyopathy in which the left ventricle (LV) of the heart does not develop properly due to impaired myocardial compaction. In utero, cardiac muscle is initially sponge-like, eventually becoming smooth and firm through a process termed compaction. Specifically, in LVNC, impairment of compaction leads to the distal portion of the LV myocardium being thicker and more sponge-like than normal. Hypertrabeculation of the myocardium, where pieces of the heart muscle extend into the LV, result in blood-filled trabeculae and intertrabecular recesses forming within the inner endocardial wall. Collectively, this impairs the LV's ability to pump oxygenated blood throughout the body.

Although various strategies are used to manage LVNC once diagnosed, the severity of comorbidities caused by LVNC, including but not limited to atrial fibrillation, embolism, or stroke, warrant further investigation into the risk factors, etiology and management of LVNC. Furthermore, patients with a definitive diagnosis of LVNC are at an elevated risk of experiencing sudden cardiac arrest (SCA) or sudden cardiac death (SCD). However, little is known about risk stratification with regards to LVNC that can result in SCA or SCD, further highlighting the need for greater analysis of the risk factors implicated in this disease state.

Ultimately, a holistic understanding of the risk factors of LVNC and subsequent morbidities it causes is needed to help improve the diagnosis, treatment and management of patients with LVNC. Hence, the goal of this study is to evaluate the risk factors and mutations associated with cardiovascular events in patients with a confirmed diagnosis of LVNC who have preserved cardiac function.

This study aims to further investigate the risk factors associated with the onset and development of LVNC. Specifically, data will be collected from retrospective and prospective patients. The retrospective cohort consists of patients who are no longer being actively followed by physicians at the Inherited Arrhythmia Clinic at the London Health Sciences Centre, University Hospital Campus, whose data will be collected annually from their medical records from the past ten years. The prospective cohort consists of patients who are being actively followed by physicians at the Inherited Arrhythmia Clinic who, once consented and enrolled, will have their charts accessed annually for the next ten years.

ELIGIBILITY:
Inclusion Criteria

Patients must meet the following criteria in order to be included in the study.

* Have a confirmed diagnosis of LVNC (between 2010-2020 for patients in the retrospective cohort only)
* Be over 18 years of age

Exclusion Criteria

Patients are ineligible to participate in this study if they do not meet one or more of the inclusion criterion or if they have any other cardiomyopathy aside from LVNC that is linked to a genetic mutation they carry.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in this study have a confirmed diagnosis of LVNC. Specifically, those in the prospective cohort are being actively followed up by physicians at the Inherited Arrhythmia Clinic whereas those in the retrospective cohort are no longer being actively followed up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2033-08-01 (Estimated); Study Completion 2033-08-01 (Estimated)

PRIMARY OUTCOMES:
Develop a large clinical registry linked with the Inherited Arrhythmia Clinic | Up to 10 years
  The Inherited Arrhythmia Clinic is a subdivision of the London Heart Rhythm Program at University Hospital, London Health Sciences Centre. As such, data will not go offsite but will simply be stored in a local REDCap database.

SECONDARY OUTCOMES:
Identification of genetic mutations linked to LVNC | Up to 10 years
  Enrolled patient's will have their genetic test results thoroughly reviewed (if applicable) to better understand their involvement in the onset and progression of LVNC.
Identification of determinants that cause LV dysfunction | Up to 10 years
  Enrolled patient's will have their medical charts accessed to identify factors contributing to LV dysfunction in patients with LVNC.
Identification of factors that lead to ICD implantation | Up to 10 years
  Enrolled patient's will have their medical charts accessed to identify risk factors that lead to ICD implantation (if applicable) in patients with LVNC.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada